CLINICAL TRIAL: NCT01480024
Title: Effect of Body Composition and Metabolism on Oocyte Gene Expression
Status: Completed | Type: Observational
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 131386
Record Dates: First submitted 2011-11-23; First posted 2011-11-28 (Estimated); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Healthy
Keywords: healthy women; oocytes; in vitro fertilization; pregnancy; childbearing-age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — oocytes and follicular fluid
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators will test the hypothesis that obese women have a unique oocyte gene expression profile that differs significantly from that of normal weight women.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 25 (N=35) or BMI ≥ 30 (N=35)
* Seeking fertility treatment at the Arkansas Fertility and Gynecology Associates Clinic
* Assisted reproduction will include the oocyte retrieval technique
* 18 to 38 years of age

Exclusion Criteria:

* Any health condition or medication that may interfere with the study outcome as determined by the investigators

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: women of childbearing age undergoing fertility treatment
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2011-04; Primary Completion 2019-05-02 (Actual); Study Completion 2019-05-02 (Actual)

PRIMARY OUTCOMES:
oocyte gene expression profile | 1-2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Arkansas Children's Nutrition Center, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] Ruebel ML, Cotter M, Sims CR, Moutos DM, Badger TM, Cleves MA, Shankar K, Andres A. Obesity Modulates Inflammation and Lipid Metabolism Oocyte Gene Expression: A Single-Cell Transcriptome Perspective. J Clin Endocrinol Metab. 2017 Jun 1;102(6):2029-2038. doi: 10.1210/jc.2016-3524. PMID 28323970